CLINICAL TRIAL: NCT05283746
Title: A Phase 1, Multicenter, Open-Label, Parallel-Group Study to Assess the Safety and Pharmacokinetics of Oral Epetraborole Tablets in Adult Subjects With Varying Degrees of Renal Function
Brief Title: A Study of Epetraborole Tablets in Subjects With Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AN2 Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EBO-102
Record Dates: First submitted 2022-02-17; First posted 2022-03-17 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): All subjects in Cohorts 1-4 receive 500 mg epetraborole once; Subjects on Cohort 5 receive 500 mg epetraborole twice
  Interventions: Drug: Epetraborole

INTERVENTIONS:
Drug: Epetraborole — Epetraborole hydrochloride 250 mg tablets for oral administration
  Other Names: AN2-501971

SUMMARY:
This is a Phase 1 study to evaluate the pharmacokinetics (PK), safety and tolerability of epetraborole tablets in adult subjects with normal renal function, subjects with various degrees of renal impairment, and subjects with end-stage renal disease (ESRD) receiving intermittent hemodialysis (IHD) therapy.

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-randomized, parallel group study in which a total of 40 subjects will be enrolled in one of 5 cohorts (8 subjects per cohort). Subjects will be enrolled based on their estimated glomerular filtration rate (eGFR) calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

* Cohort 1: Normal renal function (eGFR ≥ 90 mL/min/1.73 m2)
* Cohort 2: Mild renal impairment (eGFR ≥ 60 and < 90 mL/min/1.73 m2)
* Cohort 3: Moderate renal impairment (eGFR ≥ 30 and < 60 mL/min/1.73 m2)
* Cohort 4: Severe renal impairment (eGFR < 30 mL/min/1.73 m2)
* Cohort 5: ESRD (eGFR < 15 mL/min/1.73 m2) receiving IHD. Subjects must be stable and receiving IHD at least 3 times a week for at least 3 months prior to Screening.

ELIGIBILITY:
Inclusion Criteria:

* All subjects:

  1. Adult males or females of 18 years of age or older at the time of Screening
  2. Willing and able to provide written informed consent
  3. BMI between 18.0 and 40.0 kg/m2 (inclusive) and weight of at least 50.0 kg
  4. Have suitable venous access for blood sampling
  5. Light-, non- or ex-smoker (A light smoker is defined as someone using 10.0 nicotine units or less per day for at least 90 days prior to the first study drug administration. An ex smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
  6. Ability and willingness to abstain from alcohol from 48 hours prior to the first study drug administration until discharge from the clinical unit
  7. Be willing and able to comply with all study assessments and adhere to the protocol schedule, including the entire confinement period and the follow-up visit
  8. If female of childbearing potential, must agree to and comply with using 1 barrier method (eg, female condom or male partner using a condom) with 1 other highly effective method of birth control (eg, oral contraceptive, implant, injectable, indwelling intrauterine device, vasectomized partner), or sexual abstinence, for the duration of the study (from signing of consent to the follow-up visit) and for 30 days after last study drug administration. Females of childbearing potential must also agree not to donate ova or oocytes (ie, human eggs) during the study, and for 1 menstrual cycle after completion of the study. To be considered of non-childbearing potential, a female must have had a tubal ligation, hysterectomy, bilateral salpingo oophrectomy, or be menopaused (last menstruation >12 months prior to the first study drug administration and follicle stimulating hormone in menopausal range). Provision of written documentation is not required for female sterilization and oral confirmation is adequate.
  9. Male subjects, if sexually active with a female partner of childbearing potential, must agree to and comply with using 1 barrier method of birth control (eg, male condom) with 1 other highly effective method of birth control in their partner (eg, oral contraceptive; implant, injectable, indwelling intrauterine device), or sexual abstinence, and must not donate sperm, for the duration of the study (from signing of consent to the follow-up visit) and for 90 days after last study drug administration

     Cohort 1:
  10. Medically and hemodynamically stable without CS abnormalities at the screening visit or Day -1, based on physical examination, vital signs, 12-lead ECG, and laboratory results
  11. Normal renal function with eGFR ≥ 90 mL/min/1.73m2, calculated using the CKD-EPI equation. A 24-hour urine collection for creatinine clearance test may be conducted prior to Day -1 to confirm the healthy renal function status if, as judged by an Investigator, the result of the eGFR calculated using the CKD-EPI equation at Screening does not reflect the subject's true renal function.

      Cohorts 2 to 4:
  12. Renal impairment with eGFR ≥ 60 and < 90 mL/min/1.73m2 (Cohort 2), ≥ 30 and < 60 mL/min/1.73m2 (Cohort 3), or < 30 mL/min/1.73m2 (Cohort 4), calculated using the CKD-EPI equation.

      Cohort 5:
  13. Subjects with ESRD (eGFR < 15 mL/min/1.73m2) receiving IHD at least 3 times per week for at least 3 months at Screening.

      Cohorts 2 to 5:
  14. Medically and hemodynamically stable without CS acute or chronic illness other than renal impairment that may impact the assessment of PK and safety as assessed by the Investigator, based on physical examination, vital signs, 12-lead ECG, and laboratory results

Exclusion Criteria:

All subjects:

1. Female who is lactating or is pregnant according to the pregnancy test at Screening or prior to the first study drug administration
2. Any CS medical history or abnormal findings upon physical examination, or clinical laboratory tests, not specifically excluded in other criteria below that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject
3. QTcF interval duration > 500 msec obtained as an average from the triplicate ECGs taken at least 1 minute apart after at least 5 minutes in a semi-supine, quiet rest position at Screening or prior to the first study drug administration
4. Results of biochemistry tests for alanine aminotransferase (ALT), aspartate aminotransferase (AST), and bilirubin greater than 1.5 × the upper limit of normal (ULN) for the reference laboratory, or history of chronic liver disease, cirrhosis, or biliary disease. For subjects with Gilbert's Syndrome, the subject may be included in the study at the discretion of the Investigator if the bilirubin levels are within the range for this condition.
5. Recent history (within 6 months) of known or suspected Clostridioides difficile infection
6. History of seizure disorder except childhood history of febrile seizures
7. Positive drug/alcohol testing at Screening or prior to the first study drug administration unless the positive drug screen is due to prescription drug use that is approved by the Investigator and the Sponsor's Medical Monitor
8. Positive testing for HIV, hepatitis B surface antigen, or hepatitis C virus antibody at Screening
9. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months prior to Screening
10. History of hypersensitivity reaction or anaphylaxis to any medication, unless deemed not CS by an Investigator
11. Donation of blood or plasma within 30 days prior to the first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to the first study drug administration
12. Receipt of an investigational drug within 30 days or 5 half-lives prior to the first administration of study drug, whichever is longer
13. Any other condition or prior therapy, which, in the opinion of an Investigator, would make the volunteer unsuitable for this study, including unable to cooperate fully with the requirements of the study protocol or likely to be non-compliant with any study requirements

    Cohort 1:
14. Hemoglobin, hematocrit, white blood cell count, or platelet count less than the lower limit of normal range of the reference laboratory, unless deemed not CS by an Investigator
15. Current or anticipated concomitant medications, defined as the use of any over the counter (OTC) medications within 7 days prior to study drug administration or use of prescription medications, health supplements, and herbal remedies taken within 14 days prior to study drug administration Exceptions: Hormonal contraceptives and intermittent, as-needed acetaminophen or non-steroidal anti-inflammatory drugs (NSAIDs) for the treatment of transient headache or other minor ache/pain. Discussion between the Principal Investigator and the Sponsor's Medical Monitor is encouraged regarding the acceptability of any medications prior to study drug administration.

    Cohorts 2 to 5:
16. Hemoglobin < 10.0 g/dL, white blood cell < 3,000 cells/L, or platelet count < 100,000 cells/L
17. Current or anticipated concomitant medications with the exception of hormonal contraceptives, as-needed acetaminophen or NSAIDs for the treatment of transient, minor aches/pain, or any medication deemed essential for the management of renal impairment and the treatment of concomitant stable medical conditions as per the discretion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Characterize the PK Profile of Epetraborole and M3: Maximum Plasma Concentration | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Determination of the maximum observed plasma concentration (Cmax)
Characterize the PK Profile of Epetraborole and M3: Area Under the Plasma Concentration Versus Time Curve from Time 0 to the Last Time Point Evaluated | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Determine the area under the plasma concentration versus time curve from time 0 to the last time point evaluated (AUC0-t)
Characterize the PK Profile of Epetraborole and M3: Area Under the Plasma Concentration Versus Time Curve from Time 0 to 24 hours | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Determine the area under the plasma concentration versus time curve from time 0 to 24 hours (AUC0-24)
Characterize the PK Profile of Epetraborole and M3: Area Under the Plasma Concentration Versus Time Curve from Time 0 to Infinity | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Determine area under the drug concentration versus time curve, from time zero to infinity (AUC0-∞)
Characterize the PK Profile of Epetraborole and M3: Apparent total plasma clearance of drug | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Determine the apparent total plasma clearance of drug (CL/F)
Characterize the PK Profile of Epetraborole and M3: Time to Maximum Plasma Concentration | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Determination the time to maximum plasma concentration (Tmax)
Characterize the PK Profile of Epetraborole: Plasma from Hemodialysis Flow | Cohort 5: Day 5
  Determine the AUC from 0 to the last quantifiable concentration AUClast immediately after the end of dialysis period from inflow (arterial) line
Characterize the PK Profile of Epetraborole:Plasma from Hemodialysis Flow | Cohort 5: Day 5
  Determine the AUC from 0 to the last quantifiable concentration AUClast immediately after the end of dialysis period from inflow (venous) line
Characterize the PK Profile of Epetraborole and M3 in Urine: Cumulative drug excreted in urine over time | Cohorts 1-4: Day 1 to Day 4
  Determine the cumulative amount excreted over all time intervals (0 to T), calculated as the sum of all amounts excreted from each interval (t1-t2)
Characterize the PK Profile of Epetraborole and M3 in Urine: Unchanged drug excreted in urine during the time interval | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Determine the fraction of unchanged drug excreted in urine during the time interval (expressed in %, calculated) for parent drug only
Characterize the PK Profile of Epetraborole and M3 in Urine: Renal Clearance | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Determine renal clearance (Ae(0-t)/ AUC0-T) for parent drug only
Characterize the PK Profile of Epetraborole and M3 in Dialysate: Concentration in full dialysate | Cohort 5: Day 5
  Determine amount of drug measured in the whole dialysate volume during dialysis period
Characterize the PK Profile of Epetraborole and M3 in Urine: Dialysis clearance | Cohort 5: Day 5
  Determine the Dialysis clearance over the dialysis period
Evaluate the Incidence of Treatment Emergent Adverse Events at Baseline and Through Study Completion | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Incidence, relatedness, and severity of adverse events
Evaluate Changes in Clinical Laboratory Tests from Baseline Through Study Completion | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Incidence of changes in clinical laboratory measurements from baseline
Evaluate Change in Vital Signs from Baseline Through Study Completion | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Incidence of changes in blood pressure, pulse, respiratory rate, and temperature
Evaluate Changes in 12-lead ECG Measurements from Baseline Through Study Completion | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Incidence of changes in 12-lead ECG parameters from baseline
Evaluate Physical Examination Abnormalities from Baseline Through Study Completion | Cohorts 1-4: Day 1 to Day 4; Cohort 5: Day 1 - Day 8
  Incidence of physical exam abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly S Cruz, MD, Principal Investigator — Advanced Pharma CR LLC; Thomas C Marbury, MD, Principal Investigator — Orlando Clinical Research Center; George C Canas, MD, Principal Investigator — Nucleus Network Pty Ltd.
Locations (3):
- United States (3):
  - Advanced Pharma CR, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Nucleus Network, Saint Paul, Minnesota